CLINICAL TRIAL: NCT02084329
Title: Balance and Mild Traumatic Brain Injury: The Effect of a Weighted Compression Vest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 104865
Record Dates: First submitted 2014-03-09; First posted 2014-03-11 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-04

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Physiotherapy; Physical therapy; neurotrauma rehabilitation; Rehabilitation; Balance; Balance Confidence; concussion; Post-Concussion; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weighted Compression Vest (Experimental): Weighted Compression Vest
  Interventions: Device: Weighted Compression Vest
- Control (No Intervention)

INTERVENTIONS:
Device: Weighted Compression Vest
  Arms: Weighted Compression Vest

SUMMARY:
After a mild traumatic brain injury (mTBI) people often report balance problems. At Parkwood hospital we have noticed that balance is improved when patients with mTBI wear a weighted compression vest. This follow up pilot study looks at the immediate effects of weighted compression vests on participants with altered balance after mTBI. Participants will be recruited from the Ministry of Health Outpatient Acquired Brain Injury (ABI) Program wait list. Then each participant will perform a series of balance and walking tests under 2 conditions : 1) wearing a weighted compression vest , 2) not wearing a weighted compression vest. It will be randomized whether participants wear the vest on the first or second testing day. Participants will also be asked how confident they are about their balance and how anxious they felt performing the assessments after each testing session. We hypothesize that the weighted compression vest will improve fatigue and anxiety immediately and 24 hours after performing a complex task, and will improve static and dynamic balance, gait variability, and walking speed in patients with mTBI, during the tasks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed concussion. Symptoms persistent for more than 3 months. Self-reported balance deficits. Participants have been referred by a physician to the Outpatient ABI team at Parkwood. Participants have been screened by the ABI team and are currently awaiting treatment. No other diagnosed orthopedic injuries or significant health conditions. Able to follow instructions

Exclusion Criteria:

* Other pre-existing vestibular problems. Other diagnosed orthopedic injuries or significant health conditions that impair balance or mobility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Modified Clinical Test of Sensory Interaction on Balance(mCTSIB) | The mCTSIB will take less than 10 minutes to administer. It will be administered twice: once on intervention day 1, and once on intervention day 2 (1 week apart). The outcome measures will be administered in the same sequence each intervention day.
  The modified Clinical Test of Sensory Interaction on Balance is designed to assess how well a person uses sensory inputs (vision, vestibular, somatosensory). As well, it provides some insight into whether each of the sensory system available for balance are being used effectively. Subjects attempt to maintain balance for 30 seconds in different set conditions involving their eyes open or closed, arms across chest, and feet together or in tandem stance. Tandem stance is when one foot's heel is in front of, and in contact with the other foot's toes. The amount of time the subject can maintain balance (up to 30 seconds) is recorded in the set condition. A subject is deemed as "unable to maintain balance" if, they step out of their set condition, or if the physiotherapist deems them to be swaying too much.
The Functional Gait Assessment (FGA) | The FGA takes less then 10 minutes to administer. It will be administered twice: once on intervention day one, and once on intervention day two (one week later).
  The FGA assesses postural stability during various walking tasks. It is a 10-item gait assessment based on the Dynamic Gait Index. Each item is scored on a 4 item ordinal scale (0-3). The maximum score is 30 (normal) and the minimum score is 0 (severe impairment). The tasks have varying demands including gait with narrow base of support, gait with eyes closed, and gait while walking backwards and gait and pivot turn. The participant will perform each task, and the observer will give the participant a mark of 0-3, depending on how well the task is performed.
The Rivermead Post-Concussion Questionnaire | This outcome measure will be completed by participants prior to testing on intervention day 1 and 2
  This is a survey that the participant fills out on their own. There are 16 items, with a 5 point ordinal scale from 0-4. "0" refers to not experienced at all, and "4" refers to a severe problem. The items are all symptoms that a person with a brain injury could possibly have. There is no time limit set upon this outcome measure, as the participant completes at his/her own pace.
The 10 Metre walk test | The test will take less than 10 minutes to administer. It will be administered twice: once on intervention day 1, and once on intervention day 2 (1 week apart). The outcome measures will be administered in the same sequence each intervention day.
  The 10 Metre Walk Test asks subjects to walk 10 meters. The time it takes for the subjects to reach 6 meters is recorded (to allow for acceleration and deceleration). The test can be performed at preferred walking speed or as fast as the subject can manage. The recorder must document if the subject chose to walk at preferred vs fast speed. Three trials are done, and averaged.
Walking While Talking on a Gait Rite Mat | This will take less than 10 minutes to administer. It will be administered twice: once on intervention day 1, and once on intervention day 2 (1 week apart). The outcome measures will be administered in the same sequence each intervention day.
  Participants will ambulate 20 feet, turn around and return. Therefore each participant will walk 40 feet in total. Subjects will participate in three separate trials, in random order. The three trials include: 1-Walking 40 feet without an additional task.; 2-walking while talking (simple): walking while reciting alphabet aloud. 3; Walking while talking- complex: walking while reciting alternate letters of alphabet aloud. The scoring involves recording the time needed to complete the distance. Meanwhile, during these trials, the Gait Rite mat will record gait variability measures.

SECONDARY OUTCOMES:
Anxiety Numerical Rating Scale | Participants will be asked to rate their anxiety before, immediately after, and 24 hours after testing on days one and two.
  Participants will be asked to rate their anxiety on a scale of 0-10. "0" will be referred to as no anxiety and "10" is addressed as extreme anxiety.
Fatigue Numerical Rating Scale | Participants will be asked to rate their fatigue before, immediately after, and 24 hours after testing on days one and two.
  Participants will be asked to rate their fatigue on a scale of 0-10. "0" will be referred to as no fatigue and "10" is addressed as extreme fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon McGuire, BScPT, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Laura Graham, MPT, Principal Investigator — Western University
Locations (1):
- Parkwood Hospital- St. Joseph's Health Care, London, Ontario, Canada